CLINICAL TRIAL: NCT05812612
Title: Study on the Treatment of COVID-19 Infection by UDCA in Patients With Autoimmune Liver Disease and Its Clinical Prognosis
Brief Title: UDCA in the Treatment of COVID-19 Infection and Its Clinical Prognosis in Patients With Autoimmune Liver Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Ditan Hospital (Other)
Responsible Party: Principal Investigator, Yao Xie, Director of Department of Hepatology Division 2, Beijing Ditan Hospital, Capital Medical University, Beijing Ditan Hospital
Other Study IDs: DTXY27
Record Dates: First submitted 2023-04-10; First posted 2023-04-13 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: COVID-19 Infection
Keywords: ursodeoxycholic acid; primary biliary cholangitis; autoimmune hepatitis; COVID-19 infection
MeSH Terms: conditions — COVID-19; Liver Cirrhosis, Biliary; Hepatitis, Autoimmune | interventions — Ursodeoxycholic Acid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- COVID-19 infection in patients with autoimmune liver disease: To study the incidence of COVID-19 infection, COVID-19, disease degree and prognosis in patients with autoimmune liver disease treated with different drugs, and to explore the impact of UDCA on COVID-19 infection, disease occurrence and clinical outcome.
  Interventions: Drug: ursodeoxycholic acid

INTERVENTIONS:
Drug: ursodeoxycholic acid — To study the incidence of COVID-19 infection and COVID-19 pneumonia in patients with autoimmune liver disease treated by UDCA, and to explore the impact of UDCA on COVID-19 infection, disease occurrence and clinical outcome.
  Other Names: UDCA

SUMMARY:
This is a two-way (retrospective+prospective) cohort study of patients with primary biliary cholangitis (PBC) and autoimmune hepatitis (AIH) infected with COVID-19. Enrolled PBC and AIH patients in clinical diagnosis and treatment at Beijing Ditan Hospital affiliated with Capital Medical University from January 2021 to December 2023. After enrollment, collect the demography data of patients, the treatment information of PBC and AIH patients, the use of ursodeoxycholic acid (UDCA) and immunosuppressants, COVID-19 vaccination, COVID-19 infection and incidence, clinical symptoms, clinical biochemistry, liver imaging, lung imaging, COVID-19 nucleic acid, COVID-19 antibody, and the incidence and treatment information of COVID-19 from January 2022 to pre enrollment. After enrollment, the corresponding treatment and clinical observation of PBC and AIH were continued, and the occurrence and incidence of COVID-19 infection were observed. For patients with COVID-19 infection during the prospective observation period, COVID-19 infection, onset and treatment were observed, including clinical symptoms, signs, heart, lung imaging, COVID-19, clinical biochemistry, disease degree, virus negative, hospital stay and prognosis. To compare the difference of COVID-19 infection rate, disease severity, clinical biochemical indicators, hospital stay and prognosis between UDCA treated and non UDCA treated patients, and to study the impact of UDCA on the occurrence, incidence and prognosis of COVID-19 infection.

DETAILED DESCRIPTION:
This is a two-way (retrospective+prospective) cohort study of patients with primary biliary cholangitis (PBC) and autoimmune hepatitis (AIH) infected with COVID-19. Enrolled PBC and AIH patients in clinical diagnosis and treatment at Beijing Ditan Hospital, Capital Medical University from January 2021 to December 2023. After enrollment, the demography data of patients, the treatment information of PBC and AIH patients, the use of ursodeoxycholic acid (UDCA) and immunosuppressants, COVID-19 vaccination, COVID-19 infection and incidence, clinical symptoms, clinical biochemistry, liver imaging, lung imaging, COVID-19 nucleic acid, COVID-19 antibody, and the incidence and treatment information of COVID-19 from January 2022 to pre enrollment were collected. Meanwhile, the corresponding treatment and clinical observation of PBC and AIH were continued, and the occurrence and incidence of COVID-19 infection were observed. For patients with COVID-19 infection during the prospective observation period, COVID-19 infection, onset and treatment were observed, including clinical symptoms, signs, heart, lung imaging, COVID-19, clinical biochemistry, disease degree, virus negative, hospital stay and prognosis. This study is aim to compare the difference of COVID-19 infection rate, disease severity, clinical biochemical indicators, hospital stay and prognosis between UDCA treated and non UDCA treated patients, and to study the impact of UDCA on the occurrence, incidence and prognosis of COVID-19 infection.

ELIGIBILITY:
Inclusion Criteria:

* Autoimmune liver disease patients who have been treated with UDCA for six months or more and those who have not been treated with UDCAExclusion.

Exclusion Criteria:

* Patients with decompensated liver cirrhosis or previous history of decompensated liver cirrhosis;
* At the same time, it is associated with other viral infections, such as hepatitis A virus, hepatitis C virus, hepatitis D virus, hepatitis E virus, HIV, etc;
* Accompanied with other serious physical and mental diseases, including uncontrolled primary kidney, heart, lung, vascular, nervous, digestive, severe metabolic diseases (such as uncontrolled hyperthyroidism, diabetes, serious complications, adrenal diseases, etc.), immunodeficiency disease, and accompanied with serious infection; History of active or suspected malignant tumors or malignant tumors.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The patients with autoimmune liver disease treated with UDCA and non UDCA in Beijing Ditan Hospital affiliated to Capital Medical University from February 2022 to December 2023 were enrolled. After enrollment, the demography data of the patients were collected. From January 2022 to January 2022, the treatment information of autoimmune liver disease, the use of UDCA drugs and corticosteroids, COVID-19 vaccination, COVID-19 infection and incidence were collected. The clinical symptoms, clinical biochemistry The examination data of lung imaging examination, COVID-19 nucleic acid and COVID-19 antibody as well as other organs and functional indicators required clinically.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2023-01-30 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of COVID-19 infection | 1 year
  Patients with autoimmune liver disease infected by COVID-19 in the observation study

SECONDARY OUTCOMES:
Severity of disease after COVID-19 infection | 1 year
  Severity indicators and hospital stay after COVID-19 infection (maximum temperature, symptom relief time, nucleic acid negative conversion time)
COVID-19 nucleic acid disappearance time | 1 year
  COVID-19 nucleic acid negative conversion time
COVID-19 infection outcome | 1 year
  Clinical outcome of COVID-19 infection including improvement or death.

CONTACTS AND LOCATIONS:
Overall Officials: Rui Song, Doctor, Principal Investigator — Beijing Ditan Hospital
Locations (1):
- Department of Hepatology Division 2, Beijing Ditan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
The first stage of the study: 1. Complete the patient enrollment, demography data, autoimmune liver disease treatment, clinical efficacy related indicators, COVID-19 vaccination information, COVID-19 incidence and treatment information collection. Complete the examination and follow-up observation of the data related to UDCA and other liver protection treatments, COVID-19 infection and clinical outcomes of patients with autoimmune liver disease after enrollment. 2. Complete regular follow-up and observation of patients, and input follow-up data.
  The second stage of the study: expected to complete database entry, complete data statistics and analysis work, and publish SCI paper.
Supporting Information: Study Protocol
Time Frame: 12 months
Access Criteria: if necessary